CLINICAL TRIAL: NCT06271941
Title: Reducing Neoplasia Recurrence After Endoscopic Resection of Large Colorectal Polyps
Acronym: ABLATION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HAPC-RCT
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer; Polyp of Colon
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic Mucosal Resection (EMR)+Hybrid Argon Plasma Coagulation (h-APC) (Experimental): Standard endoscopic mucosal resection (EMR) technique will be used for the primary removal of all polyps, utilizing submucosal injection. Electrocautery snare technique will be facilitated using standard microprocessor-controlled electrocautery (e.g., ERBE VIO Endocut 3-1-6). Ablation of the margin and base of the polypectomy site will be performed using Hybrid Argon Plasma Coagulation (h-APC, Erbe Hybrid APC).
  Interventions: Procedure: Hybrid Argon Plasma Coagulation (h-APC)
- Endoscopic Mucosal Resection (EMR) + Snare tip soft coagulation (STSC) (Active Comparator): Standard endoscopic mucosal resection (EMR) technique will be used for the primary removal of all polyps, utilizing submucosal injection. Electrocautery snare technique will be facilitated using standard microprocessor-controlled electrocautery (e.g., ERBE VIO Endocut 3-1-6). Ablation of the margin of the polypectomy site will be performed using Snare tip soft coagulation (STSC).
  Interventions: Procedure: Snare tip soft coagulation (STSC)

INTERVENTIONS:
Procedure: Hybrid Argon Plasma Coagulation (h-APC) — The hybrid argon plasma coagulation (h-APC) combines an ablation technique (APC) with the option for submucosal saline injection using a high-pressure water jet. The technique allows for the lifting of dysplastic epithelium, creating a cushion under the mucosa to facilitate the ablation of larger areas more thoroughly and with higher energy settings, while posing a low risk for side effects or complications.
  Other Names: h-APC
  Arms: Endoscopic Mucosal Resection (EMR)+Hybrid Argon Plasma Coagulation (h-APC)
Procedure: Snare tip soft coagulation (STSC) — The Snare tip soft coagulation (STSC) involves using a snare to remove polyps, while simultaneously applying soft coagulation to the surrounding tissue using a specialized tip on the snare.
  Other Names: STSC
  Arms: Endoscopic Mucosal Resection (EMR) + Snare tip soft coagulation (STSC)

SUMMARY:
Large (≥20mm) colorectal polyps often harbor areas of advanced neoplasia, making them immediate colorectal cancer (CRC) precursors. Such polyps have to be completely removed to prevent CRC and to avoid surgery and/or adjuvant therapy. The laterally spreading lesions (LSLs) are removed via endoscopic mucosal resection (EMR). However, recurrence is common. New techniques for LSL resection (hybrid argon plasma coagulation (h-APC) margin and base ablation) have shown a reduction in recurrence following the interventions.

We hypothesize that performing hybrid argon plasma coagulation (h-APC) margin and base ablation during EMR of large (≥20mm) colorectal LSLs will lead to lower rates of lesion recurrence compared to Snare tip soft coagulation (STSC) margin ablation.

DETAILED DESCRIPTION:
This trial is an open-label, two-arm, parallel-group, multicenter, randomized controlled superiority trial. Patients undergoing EMR will be randomly assigned in a 1:1 ratio to undergo additional STSC margin ablation (control group and current standard of care) or h-APC ablation of the margins and base (experimental group).

Patients will be enrolled in the study before the endoscopy procedure, or in the outpatient clinic.

Eligible patients who have consented to participate in the study will be asked to take a standard colonoscopy preparation regimen before their scheduled procedure.

EMR intervention will be performed for all eligible patients with a large laterally spreading lesions (LSLs) by expert endoscopists. Only if a polyp meets inclusion criteria, the study subject will be enrolled and randomized into one of these 2 groups:

* Group 1: EMR + h-APC margin and base thermal ablation
* Group 2: EMR + STSC of the margin

The standard EMR technique will be used for the primary removal of all polyps. Submucosal injection will be used to lift the polyp from the muscularis propria. Injection will be used as per the current standard of care using a contrast agent and a lifting agent (e.g., NaCl 0.9% or Voluven). Snare electrocautery resection will be facilitated until complete visible removal of the complete polyp. Electrocautery snare technique will be facilitated using standard microprocessor-controlled electrocautery. If residual polyp tissue cannot be removed by a snare, other means such as cold snare (i.e., for small residual polyp tissue that cannot be engaged into standard snares) or avulsive methods will be used. Randomization will be performed after resection is complete and before thermal ablation. After the complete removal of the polyp, depending on the randomization group, h-APC or STSC techniques will be used for margin and base or only margin ablation of the post-EMR defect.

If multiple large polyps are found and removed, the study polyp will be marked with two tattoos 3 cm distal and 3 cm proximal to the lesion, to clearly identify the study polyp associated scar in the follow-up colonoscopy. Polyps will be sent to the pathology lab and evaluated according to standard practice by institutional pathologists. To determine the homogeneity and depth of h-APC margin ablation in the pathology lab, some ablated margins might be resected using the standard cold snare technique.

Telephone calls after 14 days following the EMR will be conducted to assess possible adverse events that occurred within the first 14 days after EMR.

Follow-up 1: Surveillance colonoscopy occurring 6 months after the EMR intervention for the assessment of recurrence (biopsy from the post-EMR site to be confirmed by pathology) following the intervention (h-APC) and the control (STSC) techniques.

Follow-up 2: Surveillance colonoscopy at 18 months (± 6 months) after the EMR intervention for the assessment of recurrence (biopsy from the post-EMR site to be confirmed by pathology) at FU1.

Patients with visible recurrence at the EMR site will undergo additional resection for complete eradication of recurrence. Patients with no visible but pathology-confirmed recurrence will be rescheduled for another colonoscopy with subsequent treatment of the post-EMR site and another follow-up colonoscopy for biopsies and confirmation of complete/incomplete eradication within 18 months after the initial EMR.

ELIGIBILITY:
Inclusion Criteria:

* adult ≥18 years old
* patients undergoing EMR for a large (≥20mm) colorectal LSL
* patients providing written and informed consent for study participation.

Exclusion Criteria:

* inflammatory bowel disease;
* non-elective colonoscopy;
* poor general health (American Society of Anesthesiologists classification >III);
* coagulopathy or thrombocytopenia (international normalized ratio ≥1.5 or platelets <50 x 109/L);
* pedunculated polyps (Paris class Ip, Isp);
* overt signs of deep submucosal invasive cancer (JNET 3);
* biopsy proven invasive carcinoma in a potential study polyp.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 892 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence after colorectal EMR between the h-APC and STSC methods | 4 years
  Lesion recurrence at first follow-up after EMR of large (≥20mm) colorectal LSLs when performing STSC margin ablation or h-APC margin and base ablation. Defined by visual recurrence or pathology-confirmed hyperplastic, serrated or adenomatous histology of the same histology of the index lesion at the tattooed resection site on at least one of four random biopsies of resection scars. These will be evaluated from an intention to treat and per protocol standpoint.

SECONDARY OUTCOMES:
Adverse event rates after EMR with STSC or h-APC | 4 years
  Adverse event rates after EMR of large (≥20mm) colorectal LSLs when performing EMR with STSC margin ablation or h-APC margin and base ablation. Defined as either a) delayed bleeding (defined as blood per rectum resulting in emergency room visit, unplanned hospitalization; endoscopic, radiologic, or surgical intervention) or b) delayed perforation (defined as endoscopic or radiologic evidence of air or luminal contents outside the gastrointestinal tract). These will be evaluated from an intention to treat and per protocol standpoint.
Technical success of STSC or h-APC | 4 years
  Technical success of STSC or h-APC defined as achieving a complete uninterrupted ring ofcircumferential margin ablation for STSC and h-APC, without crossover to complete the margin ablation, and achieving 100% surface ablation of the resection base for h-APC.
Lesion recurrence at the 18-month follow-up after EMR with STSC or h-APC | 4 years
  Lesion recurrence at the 18-month follow-up after EMR with STSC or h-APC
High-grade dysplasia or colorectal cancer occurence after EMR during the 18-month follow-up period. | 4 years
  High-grade dysplasia or colorectal cancer occurence after EMR during the 18-month follow-up period at the resection site.
CRC occurrence during the 18-month follow-up period | 4 years
  CRC occurrence after EMR during the 18-month follow-up period

OTHER OUTCOMES:
Colonoscopies required to achieve lesion clearance after EMR with STSC or h-APC | 4 years
  Colonoscopies required to achieve lesion clearance, defined as no histologic recurrence at the resection scar on follow-up.
EMR procedure time | 4 years
  EMR procedure time with STSC or h-APC
STSC or h-APC ablation time | 4 years
Loss to follow-up | 4 years
Intestinal preservation 18 months after ablation | 4 years
  Defined as no surgical resection performed.
Clinically significant delayed bleeding in the proximal colon after EMR with STSC or h-APC | 14 days
  Defined as blood per rectum resulting in emergency room visit, unplanned hospitalization; endoscopic, radiologic, or surgical intervention. Proximal defined as proximal to the splenic flexure.
Clinically significant delayed bleeding in the distal colon after EMR with STSC or h-APC | 14 days
  Defined as blood per rectum resulting in emergency room visit, unplanned hospitalization; endoscopic, radiologic, or surgical intervention. Distal defined as splenic flexure and distal.
Clinically significant delayed bleeding in the entire colon after EMR with STSC or h-APC | 14 days
  Defined as blood per rectum resulting in emergency room visit, unplanned hospitalization; endoscopic, radiologic, or surgical intervention.
Delayed perforation after EMR with STSC or h-APC | 14 days
  Delayed perforation defined as endoscopic or radiologic evidence of air or luminal contents outside the gastrointestinal tract
Any delayed bleeding after EMR | 14 days
  Any delayed bleeding after EMR, defined as blood per rectum after the procedure
Defect closure time | 4 years
Technical success for complete defect closure | 4 years
  Defined as adequate apposition of the mucosal defect margins without visible submucosal areas >3 mm along the closure line.
Costs associated with procedures | 4 years
Factors associated with recurrence after colorectal EMR between the h-APC and STSC methods | 4 years
  Lesion recurrence at first follow-up after EMR of large (≥20mm) colorectal LSLs when performing STSC margin ablation or h-APC margin and base ablation. Defined by pathology-confirmed hyperplastic, serrated or adenomatous histology of the same histology of the index lesion at the tattooed resection site on at least one of four random biopsies of resection scars. Factors such as age, sex, lesion size (20-29mm, ≥30mm; 20-39mm, ≥40mm), histology, location, difficulty (difficult defined as peri-appendiceal, on the ileocecal valve, resection previously attempted and failed by a referring endoscopist), use of epinephrine in submucosal injection, submucosal lifting solution, resection type (en bloc [i.e. in one piece] vs piecemeal), technical success, study site, endoscopist yearly EMR volume, presence of intraprocedural bleeding, utilization of adjunct resection methods, ileocecal or anus involvement, polyp histology/morphology will be evaluated.
Factors associated with adverse event rates after EMR with STSC or h-APC | 30 days
  Adverse event rates after EMR of large (≥20mm) colorectal LSLs when performing EMR with STSC margin ablation or h-APC margin and base ablation. Defined as either a) delayed bleeding (defined as blood per rectum resulting in emergency room visit, unplanned hospitalization; endoscopic, radiologic, or surgical intervention) or b) delayed perforation (defined as endoscopic or radiologic evidence of air or luminal contents outside the gastrointestinal tract). Factors such as age, sex, lesion size, morphology, histology, location, complete/incomplete/no defect closure, prophylactic vessel ablation, base ablation, anticoagulant use will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 12 months and ending 36 months following article publication.
Access Criteria: Proposals should be directed to daniel.von.renteln.med@ssss.gouv.qc.ca . To gain access, data requestors will need to sign a data access agreement